CLINICAL TRIAL: NCT00090324
Title: A 6-week, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Phase 3b Study of the Efficacy and Safety of Quetiapine Fumarate (SEROQUEL™) Immediate-release Tablets Compared With Placebo in Adolescents With Schizophrenia (Abbreviated)
Brief Title: Quetiapine Fumarate (SEROQUEL) Compared to Placebo in the Treatment of Adolescent Patients With Schizophrenia
Acronym: ANCHOR 112
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1441C00112
Record Dates: First submitted 2004-08-25; First posted 2004-08-30 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: quetiapine fumarate tablets

SUMMARY:
The purpose of this study is to demonstrate efficacy and safety of quetiapine fumarate (SEROQUEL) compared with placebo in the treatment of adolescent patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide written assent and the parents or legal guardian of the patient is able to provide written informed consent before beginning and study related procedures
* Patient has a documented clinical diagnosis of schizophrenia
* Patient's parent or legal guardian will be able to accompany the patient at each scheduled study visit

Exclusion Criteria:

* Patients (female) must not be pregnant or lactating
* Patients with a known intolerance or lack of response to previous treatment with quetiapine
* Patients who have previously participated in this study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 249 (Estimated)
Dates: Start 2004-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of Quetiapine with placebo in the treatment of schizophrenia as assessed by the PANSS total score, change from baseline to Day 42

SECONDARY OUTCOMES:
Compare the effect of Quetiapine with placebo in change from baseline to Day 42 level of functioning, evaluate aggression and hostility; evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (42):
- United States (23):
  - Research Site, Dothan, Alabama
  - Research Site, Cerritos, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Alamonte, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Newton, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Las Vegas, Nevada
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Lyndhurst, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Memphis, Tennessee
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Kirkland, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Site, Aachen, Germany
- India (2):
  - Research Site, Kanpur
  - Research Site, Lucknow
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Petaling Jaya
- Philippines (4):
  - Research Site, Davao City
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (2):
  - Research Site, Poznan
  - Research Site, Torun
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Novi Sad
- Research Site, Pretoria, South Africa
- Ukraine (3):
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Odesa

REFERENCES:
- [Derived] Findling RL, McKenna K, Earley WR, Stankowski J, Pathak S. Efficacy and safety of quetiapine in adolescents with schizophrenia investigated in a 6-week, double-blind, placebo-controlled trial. J Child Adolesc Psychopharmacol. 2012 Oct;22(5):327-42. doi: 10.1089/cap.2011.0092. PMID 23083020